CLINICAL TRIAL: NCT02677116
Title: A Phase 1, Open-Label, Dose-Escalation Study of Olaratumab as a Single Agent and in Combination With Doxorubicin, Vincristine/Irinotecan, or High-Dose Ifosfamide in Pediatric Patients With Relapsed or Refractory Solid Tumors
Brief Title: A Study of Olaratumab Alone and in Combination With Standard Chemotherapies in Children With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15841; I5B-MC-JGDN (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-01-29; First posted 2016-02-09 (Estimated); Results first posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2019-06-01

CONDITIONS: Neoplasm Metastasis
MeSH Terms: conditions — Neoplasm Metastasis | interventions — olaratumab; Doxorubicin; Vincristine; Irinotecan; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Olaratumab + Doxorubicin (Part A) (Experimental): Cycle 1: Olaratumab 15 mg/kg was administered IV Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 15 mg/kg administered IV on Days 1 and 8 and doxorubicin administered IV on Days 1 and 2. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
  Interventions: Drug: Olaratumab; Drug: Doxorubicin
- Olaratumab + Vincristine + Irinotecan (Part A) (Experimental): Cycle 1: Olaratumab 15 mg/kg was administered IV Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 15 mg/kg and vincristine administered IV on Days 1 and 8. Irinotecan administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
  Interventions: Drug: Olaratumab; Drug: Vincristine; Drug: Irinotecan
- Olaratumab + Ifosfamide (Part A) (Experimental): Cycle 1: Olaratumab 15 mg/kg was administered IV Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 15 mg/kg administered IV on Days 1 and 8 of each cycle. Ifosfamide administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
  Interventions: Drug: Olaratumab; Drug: Ifosfamide
- Olaratumab + Doxorubicin (Part B) (Experimental): Cycle 1: Olaratumab 20 mg/kg was administered IV Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 20 mg/kg administered IV on Days 1 and 8 and doxorubicin administered IV on Days 1 and 2. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
  Interventions: Drug: Olaratumab; Drug: Doxorubicin
- Olaratumab + Vincristine + Irinotecan (Part B) (Experimental): Cycle 1: Olaratumab 20 mg/kg was administered IV Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 20 mg/kg and vincristine administered IV on Days 1 and 8. Irinotecan administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
  Interventions: Drug: Olaratumab; Drug: Vincristine; Drug: Irinotecan
- Olaratumab + Ifosfamide (Part B) (Experimental): Cycle 1: Olaratumab 20 mg/kg was administered IV Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 20 mg/kg administered IV on Days 1 and 8 of each cycle. Ifosfamide administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
  Interventions: Drug: Olaratumab; Drug: Doxorubicin; Drug: Ifosfamide
- Olaratumab + Doxorubicin (Part C) (Experimental): Cycle 1 and beyond: Olaratumab 20 mg/kg administered IV on Days 1 and 8 and doxorubicin administered IV on Days 1 and 2. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
  Interventions: Drug: Olaratumab; Drug: Doxorubicin
- Olaratumab + Vincristine + Irinotecan (Part C) (Experimental): Cycle 1 and beyond: Olaratumab 20 mg/kg and vincristine administered IV on Days 1 and 8. Irinotecan administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
  Interventions: Drug: Olaratumab; Drug: Vincristine; Drug: Irinotecan
- Olaratumab + Ifosfamide (Part C) (Experimental): Cycle 1 and beyond: Olaratumab 20 mg/kg administered IV on Days 1 and 8 of each cycle. Ifosfamide administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
  Interventions: Drug: Olaratumab; Drug: Ifosfamide

INTERVENTIONS:
Drug: Olaratumab — Olaratumab administered IV.
  Other Names: LY3012207
Drug: Doxorubicin — Doxorubicin administered IV.
  Arms: Olaratumab + Doxorubicin (Part A); Olaratumab + Doxorubicin (Part B); Olaratumab + Doxorubicin (Part C); Olaratumab + Ifosfamide (Part B)
Drug: Vincristine — Vincristine administered IV.
  Arms: Olaratumab + Vincristine + Irinotecan (Part A); Olaratumab + Vincristine + Irinotecan (Part B); Olaratumab + Vincristine + Irinotecan (Part C)
Drug: Irinotecan — Irinotecan administered IV.
  Arms: Olaratumab + Vincristine + Irinotecan (Part A); Olaratumab + Vincristine + Irinotecan (Part B); Olaratumab + Vincristine + Irinotecan (Part C)
Drug: Ifosfamide — Ifosfamide administered IV.
  Arms: Olaratumab + Ifosfamide (Part A); Olaratumab + Ifosfamide (Part B); Olaratumab + Ifosfamide (Part C)

SUMMARY:
The main purpose of this study is to evaluate the safety of different doses of olaratumab and to determine which dose should be used for future pediatric studies. The present study is open to children with advanced cancer or cancer that has spread to another part of the body. The study has three parts. In the first two parts, a specific dose of olaratumab will be given in 21 day cycles, followed by one of three standard chemotherapy regimens. In the third part, a specific dose of olaratumab will be given with one of three standard chemotherapy regimens in 21 day cycles. Participants will only enroll in one part.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have histological or cytological evidence of a diagnosis of solid tumor, excluding lymphomas and melanoma, but including central nervous system (CNS) tumors, that is relapsed or refractory, not be amenable to curative treatment.
* The participant has the presence of measurable and/or nonmeasurable but evaluable disease as defined by the Response Evaluation Criteria In Solid Tumors (RECIST Version 1.1). Response Assessment in Neuro-Oncology (RANO) Criteria or Macdonald Criteria should be used for CNS tumors.
* The participant has a Lansky (<16 years of age) or Karnofsky (≥16 years of age) performance score of at least 50.
* The participant has adequate hematologic, organ, and coagulation function ≤2 weeks (14 days) prior to first dose of study drug:

  * Absolute neutrophil count (ANC) ≥750 cubic millimeters (mm³)
  * Platelets ≥75,000/mm³
  * Hemoglobin ≥8 grams per deciliter (g/dL)
  * Total bilirubin (sum of conjugated + unconjugated) ≤1.5 x upper limit of normal (ULN) for age
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 x ULN
  * Serum creatinine is based on age/gender
  * Adequate coagulation function as defined by International Normalized Ratio ≤1.5 or prothrombin time ≤1.5 x ULN, and partial thromboplastin time ≤1.5 x ULN
* Both female and male participants of child-bearing potential must agree to use highly effective contraceptive precautions during the trial and up to 3 months following the last dose of olaratumab, or longer for other study drugs according to their label.
* Participants must have fully recovered from the acute toxic effects of all prior anticancer therapies or must adhere to post-treatment conditions as follows:

  * Myelosuppressive chemotherapy
  * Hematopoietic growth factors
  * Biologic (anti-neoplastic agent)
  * Antibody therapy
  * Radiation
  * Stem cell infusion without traumatic brain injury
  * Corticosteroids

Exclusion Criteria:

* Have received treatment within 21 days of the initial dose of olaratumab with an investigational product or non-approved use of a drug or device or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Participants that have had bone marrow or solid organ transplant are excluded.
* The participant has an active fungal, bacterial, and/or known severe viral infection including human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis (screening is not required).
* Female participants who are pregnant or breastfeeding are excluded.
* If the participant is to be enrolled in the doxorubicin combination arm, a left ventricular dysfunction (LVEF < 50%) or shortening fraction of <27% by echocardiogram (either multigated acquisition [MUGA] or echocardiogram [ECHO] are required, not both).
* Participants that have received prior anthracycline therapy if the participant is to be enrolled in the doxorubicin combination arm.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- United States (20):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - The Children's Hospital for Cancer and Blood Disorders, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Riley Hosptial for Children, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - St Jude Childrens Research Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Texas Childrens Hospital, Houston, Texas
  - Primary Childrens Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital Research Foundation, Seattle, Washington
- National Cancer Center Hospital, Chuo-Ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about this study: A Study of Olaratumab Alone and in Combination With Standard Chemotherapies in Children With Cancer — http://www.lillytrialguide.com/en-US/studies/pediatric-neoplasm%20metastasis/JGDN#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers include the participants who died due to any cause or disease progression, alive and on study at conclusion, but off treatment.
Groups:
- Olaratumab + Vincristine + Irinotecan (Part A): Cycle 1: Olaratumab 15 milligram/kilogram (mg/kg) was administered alone intravenously (IV) on Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 15 mg/kg and vincristine administered IV on Days 1 and 8. Irinotecan administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab + Doxorubicin (Part A): Cycle 1: Olaratumab 15 mg/kg was administered alone IV on Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 15 mg/kg administered IV on Days 1 and 8 and doxorubicin administered IV on Days 1 and 2. . Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab + Ifosfamide (Part A): Cycle 1: Olaratumab 15 mg/kg was administered alone IV on Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 15 mg/kg administered IV on Days 1 and 8 of each cycle. Ifosfamide administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab + Vincristine + Irinotecan (Part B): Cycle 1: Olaratumab 20 mg/kg was administered alone IV on Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 20 mg/kg and vincristine administered IV on Days 1 and 8. Irinotecan administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab + Doxorubicin (Part B): Cycle 1: Olaratumab 20 mg/kg was administered alone IV on Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 20 mg/kg administered IV on Days 1 and 8 and doxorubicin administered IV on Days 1 and 2. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab + Ifosfamide (Part B): Cycle 1: Olaratumab 20 mg/kg was administered alone IV on Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 20 mg/kg administered IV on Days 1 and 8 of each cycle. Ifosfamide administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
Period: Overall Study
Arm/Group | Olaratumab + Vincristine + Irinotecan (Part A) | Olaratumab + Doxorubicin (Part A) | Olaratumab + Ifosfamide (Part A) | Olaratumab + Vincristine + Irinotecan (Part B) | Olaratumab + Doxorubicin (Part B) | Olaratumab + Ifosfamide (Part B) | Olaratumab + Vincristine + Irinotecan (Part C) | Olaratumab + Ifosfamide (Part C) | Olaratumab + Doxorubicin (Part C)
Started | 10 | 11 | 9 | 10 | 1 | 13 | 6 | 4 | 4
Cycle 1 Olaratumab Alone | 10 | 11 | 9 | 10 | 1 | 13 | 6 | 4 | 4
Progressive Disease | 7 | 7 | 6 | 7 | 0 | 9 | 2 | 2 | 2
Completed | 7 | 7 | 6 | 7 | 0 | 9 | 2 | 2 | 2
Not Completed | 3 | 4 | 3 | 3 | 1 | 4 | 4 | 2 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 3 | 2 | 1 | 3 | 1 | 1 | 2
Not completed — Withdrawal by parent or guardian | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Olaratumab + Doxorubicin (Part A): Cycle 1: Olaratumab 15 mg/kg was administered alone IV on Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 15 mg/kg administered IV on Days 1 and 8 and doxorubicin administered IV on Days 1 and 2. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab + Ifosfamide (Part A): Cycle 1: Olaratumab 15 mg/kg was administered alone IV on Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 15mg/kg administered IV on Days 1 and 8 of each cycle. Ifosfamide administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab + Ifosfamide (Part B): Cycle1: Olaratumab 20 mg/kg was administered alone IV on Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 20 mg/kg administered IV on Days 1 and 8 of each cycle. Ifosfamide administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab + Ifosfamide (Part C): Cycle 1 and beyond: Olaratumab 20 mg/kg administered IV on Days 1 and 8 of each cycle. Ifosfamide administered IV on Days 1 though 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Total: Total of all reporting groups
Arm/Group | Olaratumab + Vincristine + Irinotecan (Part A) | Olaratumab + Doxorubicin (Part A) | Olaratumab + Ifosfamide (Part A) | Olaratumab + Vincristine + Irinotecan (Part B) | Olaratumab + Doxorubicin (Part B) | Olaratumab + Ifosfamide (Part B) | Olaratumab + Vincristine + Irinotecan (Part C) | Olaratumab + Ifosfamide (Part C) | Olaratumab + Doxorubicin (Part C) | Total
Number analyzed (Participants) | 10 | 11 | 9 | 10 | 1 | 13 | 6 | 4 | 4 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (5.5) | 6.8 (4.3) | 10.7 (4.3) | 10.6 (4.9) | NA (NA) — Individual value reported = 10.0. Mean and Standard Deviation were not calculated. | 12.5 (3.8) | 9.7 (5.4) | 8.0 (7.0) | 10.8 (5.1) | 10.0 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 6 | 0 | 6 | 4 | 1 | 2 | 28
  Male | 6 | 8 | 7 | 4 | 1 | 7 | 2 | 3 | 2 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 3 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 8
  White | 9 | 8 | 5 | 7 | 1 | 11 | 3 | 1 | 1 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 1 | 1 | 0 | 3 | 2 | 1 | 1 | 14
  Not Hispanic or Latino | 9 | 7 | 7 | 8 | 1 | 10 | 1 | 0 | 0 | 43
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4
  Missing | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 1 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 11 | 9 | 10 | 1 | 13 | 3 | 1 | 1 | 59
  Japan | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Olaratumab Dose Limiting Toxicities (DLTs)
Description: A dose limiting toxicity (DLT) was defined as an adverse event (AE) during the first 21 days that was possibly related to the study drug and fulfilled any of the following criteria using the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0: CTCAE Grade 3 nonhematologic toxicity, grade 4 neutropenia that lasted longer than 2 weeks, grade ≥3 thrombocytopenia complicated by hemorrhage, and any hematologic toxicity that caused a cycle delay of >14 days.
Time Frame: Parts A and B: Cycle 1 through Cycle 2 in each arm (21-day cycle); Part C: Cycle 1 only (21-day cycle)
Population: All participants who received at least one dose of study drug and had DLTs.
Measure: Count of Participants; unit: Participants
Groups:
- Olaratumab + Vincristine + Irinotecan (Part A): Cycle 1: Olaratumab 15 mg/kg was administered alone IV on Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 15 mg/kg and vincristine administered IV on Days 1 and 8. Irinotecan administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab + Doxorubicin (Part A): Cycle 1: Olaratumab 15 mg/kg was administered alone IV on Days 1 and 8).
  Cycle 2 and beyond: Olaratumab 15 mg/kg administered IV on Days 1 and 8 and doxorubicin administered IV on Days 1 and 2. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab + Ifosfamide (Part B): Cycle 1: Olaratumab 20 mg/kg alone (administered IV on Days 1 and 8).
  Cycle 2 and beyond: Olaratumab 20 mg/kg administered IV on Days 1 and 8 of each cycle. Ifosfamide administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
Arm/Group | Olaratumab + Vincristine + Irinotecan (Part A) | Olaratumab + Ifosfamide (Part A) | Olaratumab + Doxorubicin (Part A) | Olaratumab + Vincristine + Irinotecan (Part B) | Olaratumab + Ifosfamide (Part B) | Olaratumab + Doxorubicin (Part B) | Olaratumab + Vincristine + Irinotecan (Part C) | Olaratumab + Ifosfamide (Part C) | Olaratumab + Doxorubicin (Part C)
Number analyzed (Participants) | 10 | 9 | 11 | 10 | 13 | 1 | 6 | 4 | 4
Participants | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Olaratumab Part A
Description: Pharmacokinetics (PK): Maximum serum concentration (Cmax) data of Olaratumab was reported from available sample data.
Time Frame: Cycle 1, Day 8 and Cycle 2, Days 1 and 8: 1.25 hour (h), 2.5 h, 3.5h Postdose
Population: All participants who had evaluable PK individual serum concentration samples analyzed for Cycle 1 Olaratumab alone and Cycle 2 Olaratumab combinations for Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (μg/mL)
Groups:
- Olaratumab Alone (Part A): Cycle 1: Olaratumab 15 mg/kg was administered alone IV on Days 1 and 8.
  All cycles are 21 days.
- Olaratumab + Doxorubicin (Part A): Cycle 2 and beyond: Olaratumab 15 mg/kg administered IV on Days 1 and 8. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab + Ifosfamide (Part A): Cycle 2 and beyond: Olaratumab 15 mg/kg administered IV on Days 1 and 8 of each cycle. Ifosfamide administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab + Vincristine + Irinotecan (Part A): Cycle 2 and beyond: Olaratumab 15 mg/kg and vincristine administered IV on Days 1 and 8. Irinotecan administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
Arm/Group | Olaratumab Alone (Part A) | Olaratumab + Doxorubicin (Part A) | Olaratumab + Ifosfamide (Part A) | Olaratumab + Vincristine + Irinotecan (Part A)
Number analyzed (Participants) | 28 | 6 | 9 | 7
microgram/milliliter (μg/mL)
  Cycle 1, Day 8: number analyzed (Participants) | 28 | 0 | 0 | 0
  Cycle 1, Day 8 | 439 (23) |  |  |
  Cycle 2, Day 1: number analyzed (Participants) | 0 | 6 | 9 | 7
  Cycle 2, Day 1 |  | 406 (21) | 396 (39) | 437 (44)
  Cycle 2, Day 8: number analyzed (Participants) | 0 | 6 | 8 | 6
  Cycle 2, Day 8 |  | 422 (30) | 398 (44) | 523 (26)

3. Secondary Outcome: PK: Maximum Concentration (Cmax) of Olaratumab Part B
Description: PK: Maximum serum concentration (Cmax) data of Olaratumab was reported from available sample data.
Time Frame: Cycle 1, Day 8 and Cycle 2, Days 1 and 8: 1.25 hour (h), 2.5 h, 3.5h Postdose
Population: All participants who had evaluable PK individual serum concentration samples analyzed for Cycle 1 Olaratumab alone and Cycle 2 Olaratumab combinations for Part B. Zero participants analyzed for Olaratumab and Doxorubicin being below the quantifiable limit.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (μg/mL)
Groups:
- Olaratumab Alone (Part B): Cycle 1: Olaratumab 20-mg/kg was administered alone IV on Days 1 and 8.
  All cycles are 21 days.
- Olaratumab + Doxorubicin (Part B): Cycle 2 and beyond: Olaratumab 20 mg/kg administered IV on Days 1 and 8 and doxorubicin administered IV on Days 1 and 2. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab + Ifosfamide (Part B): Cycle 2 and beyond: Olaratumab 20 mg/kg administered IV on Days 1 and 8 of each cycle. Ifosfamide administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab +Vincristine + Irinotecan (Part B): Cycle 2 and beyond: Olaratumab 20 mg/kg and vincristine administered IV on Days 1 and 8. Irinotecan administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
Arm/Group | Olaratumab Alone (Part B) | Olaratumab + Doxorubicin (Part B) | Olaratumab + Ifosfamide (Part B) | Olaratumab +Vincristine + Irinotecan (Part B)
Number analyzed (Participants) | 21 | 0 | 11 | 8
microgram/milliliter (μg/mL)
  Cycle 1, Day 8: number analyzed (Participants) | 21 | 0 | 0 | 0
  Cycle 1, Day 8 | 639 (27) |  |  |
  Cycle 2, Day 1: number analyzed (Participants) | 0 | 0 | 11 | 7
  Cycle 2, Day 1 |  |  | 629 (32) | 585 (30)
  Cycle 2, Day 8: number analyzed (Participants) | 0 | 0 | 11 | 8
  Cycle 2, Day 8 |  |  | 696 (27) | 647 (27)

4. Secondary Outcome: PK: Maximum Concentration (Cmax) of Olaratumab Part C
Description: Pharmacokinetics (PK): Maximum serum concentration (Cmax) data of Olaratumab was reported from available sample data.
Time Frame: Cycle 1, Days 1 and 8; Cycle 2, Days 1 and 8: 1.25 hour (h), 2.5 h, 3.5h Postdose
Population: All participants who had evaluable PK individual serum concentration samples analyzed for Cycle 1 and 2 for all Part C treatment combinations. Per protocol, the Part C olaratumab alone was not collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (μg/mL)
Groups:
- Olaratumab + Doxorubicin Cycle 1 (Part C): Cycle 1: Olaratumab 20 mg/kg administered IV on Days 1 and 8 and doxorubicin administered IV on Days 1 and 2. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab + Doxorubicin (Part C): Cycle 2 and beyond: Olaratumab 20 mg/kg administered IV on Days 1 and 8 and doxorubicin administered IV on Days 1 and 2. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
Arm/Group | Olaratumab + Doxorubicin Cycle 1 (Part C) | Olaratumab + Doxorubicin (Part C) | Olaratumab + Vincristine + Irinotecan (Part C) | Olaratumab + Ifosfamide (Part C)
Number analyzed (Participants) | 4 | 3 | 6 | 4
microgram/milliliter (μg/mL)
  Cycle 1, Day 1: number analyzed (Participants) | 4 | 0 | 5 | 4
  Cycle 1, Day 1 | 406 (20) |  | 548 (15) | 363 (39)
  Cycle 1, Day 8: number analyzed (Participants) | 3 | 0 | 6 | 4
  Cycle 1, Day 8 | 493 (20) |  | 695 (37) | 498 (43)
  Cycle 2, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0
  Cycle 2, Day 8: number analyzed (Participants) | 0 | 3 | 4 | 3
  Cycle 2, Day 8 |  | 502 (38) | 707 (3) | 567 (38)

5. Secondary Outcome: PK: Trough Serum Minimum Concentration (Cmin) of Olaratumab Part A
Description: PK: Trough serum concentration (Cmin) of Olaratumab was reported. A sample was collected every other cycle from cycles 1, 2, 3-25.
Time Frame: Cycles 1, 2, 3-25; Day 8: 336 Hours Postdose
Population: All participants who had evaluable PK individual serum concentration samples analyzed for Cycle 1 Olaratumab alone and Cycle 2 and 3-25 Olaratumab combinations for Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Olaratumab Alone (Part A) | Olaratumab + Doxorubicin (Part A) | Olaratumab + Ifosfamide (Part A) | Olaratumab + Vincristine + Irinotecan (Part A)
Number analyzed (Participants) | 6 | 5 | 9 | 17
μg/mL
  Cycle 1, Day 8: number analyzed (Participants) | 6 | 0 | 9 | 7
  Cycle 1, Day 8 | 73 (56) |  | 46.3 (284) | 97.8 (29)
  Cycle 2, Day 8: number analyzed (Participants) | 0 | 3 | 3 | 3
  Cycle 2, Day 8 |  | 38.5 (29.1) | 114 (85) | 37.7 (112)
  Cycle 3-25, Day 8: number analyzed (Participants) | 0 | 5 | 5 | 17
  Cycle 3-25, Day 8 |  | 94.4 (41) | 88.2 (77) | 95.1 (85)

6. Secondary Outcome: PK: Trough Serum Minimum Concentration (Cmin) of Olaratumab Part B
Description: as for outcome 5
Time Frame: Cycles 1, 2, 3-25; Day 8: 336 Hours Postdose
Population: All participants who had evaluable PK individual serum concentration samples analyzed for Cycle 1, 2 and Cycle 3-25 Olaratumab combinations for Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Olaratumab Alone (Part B): Cycle 1: Olaratumab 20 mg/kg was administered alone IV on Days 1 and 8.
  All cycles = 21 days
- Olaratumab +Vincristine + Irinotecan (Part B): Cycle 1: Olaratumab 20 mg/kg was administered alone IV on Days 1 and 8.
  Cycle 2 and beyond: Olaratumab 20 mg/kg and vincristine administered IV on Days 1 and 8. Irinotecan administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
Arm/Group | Olaratumab Alone (Part B) | Olaratumab + Doxorubicin (Part B) | Olaratumab + Ifosfamide (Part B) | Olaratumab +Vincristine + Irinotecan (Part B)
Number analyzed (Participants) | 0 | 0 | 11 | 9
μg/mL
  Cycle 1, Day 8 |  |  | 125 (55) | 99.1 (65)
  Cycle 2, Day 8: number analyzed (Participants) | 0 | 0 | 4 | 3
  Cycle 2, Day 8 |  |  | 199 (36) | 230 (17)
  Cycle 3-25, Day 8: number analyzed (Participants) | 0 | 0 | 5 | 6
  Cycle 3-25, Day 8 |  |  | 289 (14) | 348 (15)

7. Secondary Outcome: PK: Trough Serum Minimum Concentration (Cmin) of Olaratumab Part C
Description: as for outcome 5
Time Frame: Cycles 1, 2, 3-25; Day 8: 336 Hours Postdose
Population: All participants who had evaluable PK individual serum concentration samples analyzed for Cycle 1, 2 and Cycle 3-25 Olaratumab combinations for Part C.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Olaratumab + Doxorubicin (Part C) | Olaratumab + Vincristine + Irinotecan (Part C) | Olaratumab + Ifosfamide (Part C)
Number analyzed (Participants) | 3 | 5 | 3
μg/mL
  Cycle 1, Day 8 | 90.3 (33) | 83.7 (8) | 124 (32)
  Cycle 2, Day 8: number analyzed (Participants) | 2 | 3 | 1
  Cycle 2, Day 8 | 141 (18) | 134 (54) | NA (NA) — Geometric mean and geometric coefficient of variation (CV) was not calculated due to one participant; individual participant data reported: 250.
  Cycle 3-25, Day 8: number analyzed (Participants) | 2 | 3 | 1
  Cycle 3-25, Day 8 | 156 (24) | 83.7 (48) | NA (NA) — Geometric mean and geometric coefficient of variation (CV) was not calculated due to one participant; individual participant data reported: 210.

8. Secondary Outcome: Percentage of Participants With a Complete Response (CR) or Partial Response (PR) (Objective Response Rate [ORR])
Description: Objective Response Rate (ORR) is the percentage of participants achieving a confirmed best overall tumor response of CR or PR. According to RECIST v1.1, PR defined as a >30% decrease in the sum of the longest diameters (LD) of the target lesions, taking as reference the baseline sum of the LD; CR was defined as the disappearance of all target and non-target lesions.
Time Frame: Baseline to objective progression or start of new anti-cancer therapy (Up to 7 months)
Population: All participants who received at least one dose of study drug and had evaluable ORR data.
Measure: Number; unit: percentage of participants
Groups:
- Olaratumab + Ifosfamide (Part B): Cycle 1: Olaratumab 20 mg/kg was administered alone IV on Days 1 and 8.
  Cycle 2 and beyond: Olaratumab administered IV on Days 1 and 8 of each cycle. Ifosfamide administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
Arm/Group | Olaratumab + Vincristine + Irinotecan (Part A) | Olaratumab + Ifosfamide (Part A) | Olaratumab + Doxorubicin (Part A) | Olaratumab + Vincristine + Irinotecan (Part B) | Olaratumab + Ifosfamide (Part B) | Olaratumab + Doxorubicin (Part B) | Olaratumab + Vincristine + Irinotecan (Part C) | Olaratumab + Ifosfamide (Part C) | Olaratumab + Doxorubicin (Part C)
Number analyzed (Participants) | 10 | 9 | 11 | 10 | 13 | 1 | 6 | 4 | 4
percentage of participants | 0 | 0 | 9.1 | 20.0 | 0 | 0 | 0 | 0 | 25.0

9. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from baseline to the first date of radiological disease progression or death due to any cause. Progressive disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). The appearance of one or more new lesions is also considered progression. If participant started new treatment before PD, the participant was censored at the date of last tumor assessment prior to new therapy. If treatment was discontinued for reasons other than PD and no further assessment, censoring occurred at last tumor assessment.
Time Frame: Baseline to radiological disease progression or death from any cause (Up to 2 Years)
Population: All participants who received at least one dose of study drug. Censored participants: Parts A-C include arms: Olaratumab + Vincristine + Irinotecan, Olaratumab + Ifosfamide and Olaratumab + Doxorubicin. Part A censored participants are 2, 2, and 2; Part B censored participants are 2, 2, and 1 and Part C censored participants are 2,1, and 4.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Olaratumab + Ifosfamide (Part B): Cycle 1: Olaratumab 20 mg/kg was administered alone IV on Days 1 and 8.
  Cycle 2 and beyond: Olaratumab administered IV on Days 1 and 8 of each cycle. Ifosfamide administered IV on Days 1 though 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
Arm/Group | Olaratumab + Vincristine + Irinotecan (Part A) | Olaratumab + Ifosfamide (Part A) | Olaratumab + Doxorubicin (Part A) | Olaratumab + Vincristine + Irinotecan (Part B) | Olaratumab + Ifosfamide (Part B) | Olaratumab + Doxorubicin (Part B) | Olaratumab + Vincristine + Irinotecan (Part C) | Olaratumab + Ifosfamide (Part C) | Olaratumab + Doxorubicin (Part C)
Number analyzed (Participants) | 10 | 9 | 11 | 10 | 13 | 1 | 6 | 4 | 4
Months | 1.54 [0.69 to 15.74] | 1.38 [0.62 to 5.68] | 1.26 [0.26 to 5.26] | 1.28 [0.53 to 11.07] | 1.25 [1.15 to 3.12] | NA [NA to NA] — The PFS was not calculated for median and 95% confidence interval due to n=1. | 4.07 [1.41 to 4.07] | 4.88 [0.69 to 8.54] | 5.52 [1.22 to 5.52]

10. Secondary Outcome: Percentage of Participants With Treatment Emergent (TE) Positive Anti-Olaratumab Antibodies
Description: Percentage of participants with a TE positive anti-olaratumab antibodies defined as a participant with a 4-fold (2 dilutions) increase over a positive baseline antibody titer.
Time Frame: From Baseline to Study Completion (Up to 33 Months)
Population: All participants who received at least one dose of study drug and had evaluable baseline sample and at least 1 evaluable post baseline sample.
Measure: Number; unit: percentage of participants
Arm/Group | Olaratumab + Vincristine + Irinotecan (Part A) | Olaratumab + Ifosfamide (Part A) | Olaratumab + Doxorubicin (Part A) | Olaratumab + Vincristine + Irinotecan (Part B) | Olaratumab + Ifosfamide (Part B) | Olaratumab + Doxorubicin (Part B) | Olaratumab + Vincristine + Irinotecan (Part C) | Olaratumab + Ifosfamide (Part C) | Olaratumab + Doxorubicin (Part C)
Number analyzed (Participants) | 10 | 9 | 11 | 10 | 13 | 1 | 6 | 4 | 4
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 33 Months.
Description: All participants who received at least one dose of study drug up to 30 days after last dose of study drug. Gender specific events only occurring in male and female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Olaratumab + Vincristine + Irinotecan (Part B): Cycle 1: Olaratumab 20 mg/kg administered alone IV on Days 1 and 8. Cycle 2 and beyond: Olaratumab 20 mg/kg and vincristine administered IV on Days 1 and 8. Irinotecan administered IV on Days 1 through 5. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
- Olaratumab + Doxorubicin (Part B): Cycle 1: Olaratumab 20 mg/kg alone was administered alone IV on Days 1 and 8. Cycle 2 and beyond: Olaratumab 20 mg/kg administered IV on Days 1 and 8 and doxorubicin administered IV on Days 1 and 2. Treatment will cease when discontinuation criterion is met.
  All cycles are 21 days.
Arm/Group | Olaratumab + Vincristine + Irinotecan (Part A) | Olaratumab + Ifosfamide (Part A) | Olaratumab + Doxorubicin (Part A) | Olaratumab + Vincristine + Irinotecan (Part B) | Olaratumab + Ifosfamide (Part B) | Olaratumab + Doxorubicin (Part B) | Olaratumab + Vincristine + Irinotecan (Part C) | Olaratumab + Ifosfamide (Part C) | Olaratumab + Doxorubicin (Part C)
All-Cause Mortality (participants affected / at risk) | 2/10 | 1/9 | 2/11 | 2/10 | 2/13 | 0/1 | 0/6 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 3/10 | 4/9 | 2/11 | 5/10 | 7/13 | 0/1 | 2/6 | 1/4 | 4/4
Other Adverse Events (participants affected / at risk) | 10/10 | 9/9 | 11/11 | 9/10 | 13/13 | 1/1 | 6/6 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Olaratumab + Vincristine + Irinotecan (Part A) (N=10) | Olaratumab + Ifosfamide (Part A) (N=9) | Olaratumab + Doxorubicin (Part A) (N=11) | Olaratumab + Vincristine + Irinotecan (Part B) (N=10) | Olaratumab + Ifosfamide (Part B) (N=13) | Olaratumab + Doxorubicin (Part B) (N=1) | Olaratumab + Vincristine + Irinotecan (Part C) (N=6) | Olaratumab + Ifosfamide (Part C) (N=4) | Olaratumab + Doxorubicin (Part C) (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 6 (8) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile infection (Infections and infestations) | 0/6 (0) | 1/7 (1) | 0/8 (0) | 0/4 (0) | 0/7 (0) | 0 (0) | 0/2 (0) | 0/3 (0) | 0/2 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shunt occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaratumab + Vincristine + Irinotecan (Part A) (N=10) | Olaratumab + Ifosfamide (Part A) (N=9) | Olaratumab + Doxorubicin (Part A) (N=11) | Olaratumab + Vincristine + Irinotecan (Part B) (N=10) | Olaratumab + Ifosfamide (Part B) (N=13) | Olaratumab + Doxorubicin (Part B) (N=1) | Olaratumab + Vincristine + Irinotecan (Part C) (N=6) | Olaratumab + Ifosfamide (Part C) (N=4) | Olaratumab + Doxorubicin (Part C) (N=4)
Anaemia (Blood and lymphatic system disorders) | 4 (9) | 7 (36) | 6 (11) | 5 (18) | 8 (55) | 0 (0) | 4 (12) | 3 (5) | 4 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (7) | 0 (0) | 0 (0) | 2 (16) | 2 (9) | 0 (0) | 3 (21) | 2 (16) | 3 (23)
Lymphopenia (Blood and lymphatic system disorders) | 1 (6) | 0 (0) | 0 (0) | 1 (7) | 2 (7) | 0 (0) | 0 (0) | 2 (6) | 3 (26)
Neutropenia (Blood and lymphatic system disorders) | 1 (8) | 0 (0) | 1 (1) | 2 (26) | 2 (8) | 0 (0) | 4 (19) | 2 (13) | 3 (24)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (16) | 0 (0) | 0 (0) | 1 (7) | 3 (14) | 0 (0) | 2 (3) | 0 (0) | 3 (15)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (8) | 1 (2) | 1 (7) | 1 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling of eyelid (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (9) | 0 (0) | 1 (1) | 5 (10) | 2 (2) | 0 (0) | 2 (6) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (6) | 1 (1) | 3 (6) | 2 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (41) | 1 (1) | 1 (1) | 7 (20) | 1 (1) | 0 (0) | 6 (21) | 2 (6) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (31) | 4 (12) | 4 (5) | 7 (24) | 9 (34) | 1 (1) | 2 (4) | 3 (10) | 3 (5)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (4) | 2 (6) | 0 (0) | 0 (0) | 2 (3) | 1 (6)
Vomiting (Gastrointestinal disorders) | 7 (34) | 5 (17) | 4 (8) | 5 (14) | 8 (11) | 0 (0) | 3 (4) | 2 (7) | 2 (4)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 6 (15) | 2 (3) | 4 (4) | 3 (6) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (4) | 3 (3) | 4 (10) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Recall phenomenon (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (9) | 2 (9) | 1 (1) | 1 (3) | 2 (3) | 1 (1) | 3 (7) | 2 (8) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 4 (6) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 3 (4) | 2 (7) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 2 (3) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram pr shortened (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophil percentage decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 (0)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (3) | 5 (29) | 2 (6) | 3 (4) | 0 (0) | 0 (0) | 2 (11) | 1 (11) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (16) | 3 (13) | 5 (22) | 3 (4) | 3 (4) | 0 (0) | 1 (3) | 2 (9) | 1 (7)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ph urine increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 7 (43) | 3 (12) | 1 (2) | 5 (30) | 0 (0) | 3 (11) | 1 (8) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 2 (15) | 7 (45) | 3 (21) | 3 (8) | 4 (16) | 0 (0) | 1 (2) | 2 (13) | 1 (6)
White blood cell count increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (8) | 1 (2) | 2 (2) | 2 (3) | 3 (5) | 0 (0) | 2 (5) | 2 (4) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (9) | 2 (10) | 0 (0) | 1 (1) | 4 (11) | 0 (0) | 1 (2) | 2 (5) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (5) | 3 (5) | 1 (1) | 2 (2) | 3 (6) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (12) | 4 (5) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (5) | 2 (8) | 0 (0) | 2 (2) | 5 (14) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 4 (5) | 1 (1) | 1 (2) | 5 (16) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 2 (2) | 3 (5) | 4 (14) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Hypouricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Refeeding syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 4 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (4) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 3 (3) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (8) | 2 (5) | 0 (0) | 6 (8) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Hemiparesis (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Writer's cramp (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fanconi syndrome acquired (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ketonuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (9) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (3) | 1 (2) | 1 (1) | 1 (2) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 2 (3) | 2 (3) | 4 (4) | 0 (0) | 3 (3) | 2 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 4 (5) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0) | 1 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT02677116/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT02677116/SAP_001.pdf